CLINICAL TRIAL: NCT07100210
Title: A Clinical Trial Evaluating the Safety, Tolerability, and Preliminary Anti-tumor Activity of IL-22BP/LNP Compound in Refractory Malignant Solid Tumors
Brief Title: A Clinical Trial Evaluating IL-22BP/LNP Compound in Refractory Malignant Solid Tumors for Safety, Tolerability and Activity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1911
Record Dates: First submitted 2024-12-08; First posted 2025-08-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Refractory Malignant Solid Tumors; mRNA Vaccine; Interleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL-22BP/LNP compound cohort (Experimental): In this study, six patients were divided into two groups (n=3 per group), which received 25 μg or 50 μg of the IL-22BP/LNP compound, respectively. The treatment will be administered by intratumoral injection. Enrolled subjects will receive inoculations of IL-22BP/LNP compound injection according to their respective dose groups, which include 5 doses for basic immunization and subsequent personalized treatment. During the basic immunization, the first 4 doses will be given at an interval of 1 week each, and the 5th dose will be administered 1 month after the 4th dose. The entire course of treatment lasts for two months.
  Interventions: Biological: IL-22BP mRNA vaccine injection

INTERVENTIONS:
Biological: IL-22BP mRNA vaccine injection — During the injection of IL-22BP/LNP compound, there were two dose groups, namely 25 μg and 50 μg of mRNA, with three participants in each dose group, aiming to evaluate the safety and tolerability of the IL-22BP/LNP compound formulation. The treatment will be administered by intratumoral injection. Enrolled subjects will receive inoculations of IL-22BP/LNP compound injection according to their respective dose groups, which include 5 doses for basic immunization and subsequent personalized treatment. During the basic immunization, the first 4 doses will be given at an interval of 1 week each, and the 5th dose will be administered 1 month after the 4th dose.The entire treatment period lasts for 2 months.

SUMMARY:
This study aims to investigate the safety and efficacy of the IL-22BP/LNP compound in patients with refractory malignant solid tumors, such as advanced soft tissue sarcoma, advanced head and neck squamous cell carcinoma, and malignant melanoma, who have failed second-line treatment, have advanced recurrence or metastatic malignant solid tumors.

DETAILED DESCRIPTION:
Cancer is a major cause of death among the global population and a significant obstacle to life extension. According to the statistics of the World Health Organization in 2019, it ranked as the first or second leading cause of death before the age of 70 in 112 countries, and in recent years, the burden of its incidence and mortality has increased rapidly. The treatment of advanced cancer consumes a large amount of resources, has poor efficacy, and is accompanied by numerous side effects. For example, the 5-year survival rate of advanced head and neck squamous cell carcinoma is only 40 - 50%, and radiotherapy may lead to osteonecrosis, while chemotherapy may cause hepatorenal toxicity and so on.

Against this background, researchers have been exploring better treatment options, and gene therapy has attracted much attention. Messenger RNA (mRNA) is a crucial part of gene therapy, and immune gene therapy holds great potential. Interleukin-22 (IL-22) influences tumor development, and IL-22 binding protein (IL-22BP) can block its activity and impede the proliferation of tumor cells.

Previously, there has been no research on mRNA vaccines targeting IL-22. Therefore, this project will provide a new treatment strategy for patients with advanced refractory malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: aged ≥ 18 years old and ≤ 70 years old;
2. Patients with histopathologically confirmed, refractory to second-line treatment, advanced recurrent/metastatic malignant solid tumors and without standard clinical treatment regimens (such as patients with advanced soft tissue sarcoma, advanced head and neck squamous cell carcinoma, malignant melanoma, etc.);
3. Eastern Cooperative Oncology Group (ECOG) performance status score: 0 - 1;
4. Expected survival time ≥ 3 months;
5. More than 28 days since the last chemotherapy/radiotherapy/surgery;
6. More than 6 weeks since the last use of nitrosoureas or mitomycin C;
7. Main organ functions are in good condition;
8. Sign a written informed consent form.

Exclusion Criteria:

1. Have participated in other drug clinical trials within 4 weeks;
2. The tumor is located close to major blood vessels or the trachea;
3. Patients with uncontrolled cardiac clinical symptoms or diseases, such as heart failure of NYHA class II or above, unstable angina pectoris, having had a myocardial infarction within 1 year, and having clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention.
4. For female subjects: pregnant or lactating women.
5. Patients have active tuberculosis, bacterial or fungal infections (≥ grade 2 of NCI-CTCAE 5.0); have active HIV infection, active HBV infection, or HCV infection.
6. Those with a history of psychotropic drug abuse who are unable to quit or have mental disorders;
7. Subjects have any active autoimmune diseases or a history of autoimmune diseases (such as, but not limited to: uveitis, enteritis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or those whose asthma in childhood has been completely relieved and who do not require any intervention in adulthood can be included; subjects with asthma that requires bronchodilators for medical intervention cannot be included).
8. Subjects are currently receiving immunosuppressive treatment.
9. Have a history of drug abuse or known medical, psychological, or social conditions, such as a history of alcoholism or drug use.
10. Known to be allergic, hypersensitive, or intolerant to the studied IL-22BP/LNP (including any excipients). Have a severe allergy history to any drugs, foods, or vaccines in the past, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, local allergic necrotizing reaction (Arthus reaction), etc.
11. From the screening period to 12 months after the completion of drug injection, female subjects have pregnancy plans or the partners of male subjects have pregnancy plans.
12. According to the investigator's judgment, there are concomitant diseases that seriously endanger patient safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities and Treatment Interruptions Due to Adverse Events During the First Cycle of IL-22BP/LNP Treatment | Participation in the whole process of the study.The entire treatment period lasts approximately 2 months.
  Evaluate the incidence of dose-limiting toxicity (DLT) during the treatment with IL-22BP/LNP compound and the number of treatment interruptions due to treatment-related adverse reactions during the first treatment cycle.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP/LNP compound was injected.The time window is approximately 2 months.
  It refers to the proportion of patients whose tumors have shrunk to a certain extent and remained so for a certain period of time. It is a direct indicator to measure the anti-tumor activity of drugs.It is usually calculated as the percentage of the sum of the number of patients with complete response (CR) and partial response (PR) in the total number of patients.
Disease Control Rate (DCR) | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP/LNP compound was injected.The time window is approximately 2 months.
  It refers to the proportion of patients whose tumors have shrunk or remained stable. It reflects the control of tumor growth by treatment, including tumor shrinkage (as involved in ORR) and the situation where the tumor does not progress.It is calculated as the percentage of the sum of the number of patients with complete response (CR), partial response (PR), and stable disease (SD) in the total number of patients.
Time to first complete remission (CR), partial remission (PR) on treatment with IL-22BP preparation. | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP/LNP compound was injected.The time window is approximately 2 months.
  Complete Response (CR): All target lesions disappear, no new lesions emerge, and tumor markers return to normal. This means that, from the perspective of imaging and relevant examinations, the tumor has completely vanished, and the patient's condition has achieved the most ideal improvement. For example, in the treatment of lymphoma, if enlarged lymph nodes completely disappear as detected by imaging examinations such as PET-CT, and relevant tumor markers in the blood also return to normal, it can be judged as a complete response.Partial Response (PR): The sum of the maximum diameters of target lesions is reduced by ≥ 30%, and no new lesions appear. Taking lung cancer as an example, if the sum of the maximum diameters of lung tumors is reduced by more than 30% after treatment and no new tumor lesions are detected, it is in a partial response state. This situation indicates that the tumor responds to the treatment and the patient's condition is under a certain degree of control.
Duration of Response(DOR) | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP/LNP compound was injected. The time window is approximately 2 months.
  DOR is defined as the time between the first confirmation of CR, PR and the first disease progression or death from any cause.
Duration of first confirmed disease stabilization | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP/LNP compound was injected.The time window is approximately 2 months.
  Defined as the time between the first confirmed stable disease (SD) and the first disease progression or death from any cause.
Progression - Free Survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Defined as the time between first treatment with IL-22BP/LNP compound and first disease progression or death from any cause progression or death from any cause.
Overall Survival(OS) | From date of randomization until the date of death from any cause, assessed up to 36 months.
  OS defined as time from first treatment with IL-22BP/LNP compound to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gersten O, Barbieri M. Evaluation of the Cancer Transition Theory in the US, Select European Nations, and Japan by Investigating Mortality of Infectious- and Noninfectious-Related Cancers, 1950-2018. JAMA Netw Open. 2021 Apr 1;4(4):e215322. doi: 10.1001/jamanetworkopen.2021.5322. PMID 33843999
- [Background] Ibarra AMC, Cecatto RB, Motta LJ, Dos Santos Franco AL, de Fatima Teixeira da Silva D, Nunes FD, Hamblin MR, Rodrigues MFSD. Photodynamic therapy for squamous cell carcinoma of the head and neck: narrative review focusing on photosensitizers. Lasers Med Sci. 2022 Apr;37(3):1441-1470. doi: 10.1007/s10103-021-03462-3. Epub 2021 Dec 2. PMID 34855034
- [Background] Sayed N, Allawadhi P, Khurana A, Singh V, Navik U, Pasumarthi SK, Khurana I, Banothu AK, Weiskirchen R, Bharani KK. Gene therapy: Comprehensive overview and therapeutic applications. Life Sci. 2022 Apr 1;294:120375. doi: 10.1016/j.lfs.2022.120375. Epub 2022 Feb 3. PMID 35123997
- [Background] Arjmand B, Larijani B, Sheikh Hosseini M, Payab M, Gilany K, Goodarzi P, Parhizkar Roudsari P, Amanollahi Baharvand M, Hoseini Mohammadi NS. The Horizon of Gene Therapy in Modern Medicine: Advances and Challenges. Adv Exp Med Biol. 2020;1247:33-64. doi: 10.1007/5584_2019_463. PMID 31845133
- [Background] Markota A, Endres S, Kobold S. Targeting interleukin-22 for cancer therapy. Hum Vaccin Immunother. 2018;14(8):2012-2015. doi: 10.1080/21645515.2018.1461300. Epub 2018 May 17. PMID 29617184
- [Background] Kempski J, Giannou AD, Riecken K, Zhao L, Steglich B, Lucke J, Garcia-Perez L, Karstens KF, Wostemeier A, Nawrocki M, Pelczar P, Witkowski M, Nilsson S, Konczalla L, Shiri AM, Kempska J, Wahib R, Brockmann L, Huber P, Gnirck AC, Turner JE, Zazara DE, Arck PC, Stein A, Simon R, Daubmann A, Meiners J, Perez D, Strowig T, Koni P, Kruglov AA, Sauter G, Izbicki JR, Guse AH, Rosch T, Lohse AW, Flavell RA, Gagliani N, Huber S. IL22BP Mediates the Antitumor Effects of Lymphotoxin Against Colorectal Tumors in Mice and Humans. Gastroenterology. 2020 Oct;159(4):1417-1430.e3. doi: 10.1053/j.gastro.2020.06.033. Epub 2020 Jun 22. PMID 32585307
- [Background] Hou X, Zaks T, Langer R, Dong Y. Lipid nanoparticles for mRNA delivery. Nat Rev Mater. 2021;6(12):1078-1094. doi: 10.1038/s41578-021-00358-0. Epub 2021 Aug 10. PMID 34394960
- [Background] Kiaie SH, Majidi Zolbanin N, Ahmadi A, Bagherifar R, Valizadeh H, Kashanchi F, Jafari R. Recent advances in mRNA-LNP therapeutics: immunological and pharmacological aspects. J Nanobiotechnology. 2022 Jun 14;20(1):276. doi: 10.1186/s12951-022-01478-7. PMID 35701851